CLINICAL TRIAL: NCT05355155
Title: An Exploratory Study of Bevacizumab Combined With FOLFOX4 in the Treatment of Recurrent Hepatocellular Carcinoma (HCC) After Liver Transplantation
Brief Title: Bevacizumab Biosimilar Plus FOLFOX4 in the Treatment of Recurrent HCC After Liver Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xuehao Wang, Head of Hepatobiliary Center；Academician of Chinese Academy of Engineering, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-SR-380
Record Dates: First submitted 2022-04-20; First posted 2022-05-02 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Post-orthotopic Liver Transplantation; Hepatocellular Carcinoma Recurrent
MeSH Terms: interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bevacizumab combine with FOLFOX4 (Experimental): Bevacizumab biosimilar：7.5mg/kg，IV，D1，Q2W FOLFOX4：
  1. Oxaliplatin: 85 mg/m2 , IV, D1，Q2W
  2. Calcium leovorin: 200 mg/m2 ,IV, D1、D2，Q2W
  3. Fluorouracil: 400 mg/m2 push infusion and given 600mg/m2 intravenously 22 hours later， D1、D2, Q2W Treatment will continue until disease progression, an unacceptable toxicity, or the patient voluntarily discontinues the study, whichever comes first.
  Interventions: Drug: Bevacizumab Biosimilar IBI305

INTERVENTIONS:
Drug: Bevacizumab Biosimilar IBI305 — Patients received bevacizumab and FOLFOX4 every two weeks
  Other Names: FOLFOX4

SUMMARY:
This study is a single arm, single center, prospective and open exploratory study.

About 15 patients with recurrent hepatocellular carcinoma (HCC) after liver transplantation are expected to be enrolled.Patients will be treated with bevacizumab and FOLFOX4.Treatment was continued until disease progression, development of intolerable toxicities, death, withdrawal of consent, initiation of new antitumor therapy, whichever occurred first.

DETAILED DESCRIPTION:
Bevacizumab biosimilar：7.5mg/kg，IV，D1，Q2W FOLFOX4：

1. Oxaliplatin: 85 mg/m2 , IV, D1，Q2W
2. Calcium leovorin: 200 mg/m2 ,IV, D1、D2，Q2W
3. Fluorouracil: 400 mg/m2 push infusion and given 600mg/m2 intravenously 22 hours later， D1、D2, Q2W

ELIGIBILITY:
Inclusion criteria:

* adult patients with hepatocellular carcinoma who have received liver transplantation have postoperative radiographic or pathological evidence of recurrence;
* have not received the first line of standard treatment or have received the first line of standard treatment failure;
* at least one measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 2;
* Child-Pugh class A or B (Child-Pugh score ≤7 );
* adequate organ function;
* a predicted life expectancy of at least 3 months.

Exclusion Criteria:

* allergy to the study drugs or their expedients or severe allergy to other monoclonal antibodies;
* receipt of attenuated inactivated vaccines within 4 weeks of the start of the study or scheduled for such vaccination during the study;
* evident concern of GI bleeding (local active ulcer, Guaic test at least ++) or a history of GI bleeding within the preceding 6 months;
* uncontrolled pleural or peritoneal effusion;
* pulmonary tuberculosis, sarcoidosis, HIV infection, or active HBV or HCV infection;
* uncontrolled cardiac arrhythmia (including QTC interval ≥500 ms);
* hepatic encephalopathy;
* Known hepatocholangiocarcinoma, mixed hepatocellular and cholangiocellular carcinoma, fibrolamellar carcinoma, or a history of or concurrent cancer except cervical carcinoma in situ and cured basal cell carcinoma;
* pregnant or lactating women or women contemplating pregnancy;
* severe concomitant illness that jeopardizes patient safety or interferes with the completion of the study as deemed by the investigators;
* esophageal or gastric variceal bleeding with portal hypertension within the past 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) ,Based on RECIST 1.1 | From the first dose of study drug to the first date of documentation of disease progression or death whichever occurred first (up to approximately 2 years )
  ORR was defined as the percentage of participants who had best overall response (BOR) of complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by investigator analysis. Responses (PR or CR) were confirmed no less than 4 weeks after the initial response. CR defined as disappearance of all target lesions and non-target lesions (a short diameter is <10 millimeter [mm] if it exists in a lymph node). PR defined as at least 30% decrease in the sum of the long diameter (LD) (hereafter referred to as sum of LD) of all target lesions, as compared with Baseline summed LD.

SECONDARY OUTCOMES:
Progression-free Survival (PFS), Based on RECIST 1.1 and mRECIST | From the first study dose date to the date of first documentation of disease progression or death (whichever occurred first) (up to approximately 2 years )
  PFS was defined as the time from the first study dose date to the date of first documentation of disease progression or death (whichever occurred first) based on RECIST 1.1 and mRECIST assessed by investigator review. PD was defined as at least a 20% increase in the sum of LD of target and non-target lesions as compared with the smallest sum of LD and the increase of LD was at least 5 mm (including new lesions).
Disease Control Rate (DCR) ,Based on RECIST 1.1 and mRECIST | Proportion of patients whose tumor volume control (reduced or enlarged) reaches a predetermined value and can maintain a minimum time limit(up to approximately 2 years)
  the proportion of patients who achieved CR, PR, or SD as their best overall response
Duration of Response (DOR) ,Based on RECIST 1.1 and mRECIST | DOR was defined as the time from the first documentation of CR or PR to the date of first documentation of PD or death (whichever occurred first) in participants with confirmed CR or PR based on RECIST 1.1 and mRECIST assessed by investigator analysis.
  From date of first documented confirmed CR or PR until date of first documentation of PD or death whichever occurred first (up to approximately 2 years)
Overall Survival (OS) | From the date of first dose of study drug until date of death from any cause (up to approximately 2 years )
  From the date of first dose of study drug until date of death from any cause (up to approximately 2 years )
Time-to Response (TTR) Based on RECIST1.1 and mRECIST | From date of first dose of study drug until CR or PR (up to approximately 2 years
  TTR was defined as the time from the date of first study dose to the date of first documentation of CR or PR, in participants with confirmed CR or PR. It was evaluated according to RECIST1.1 and mRECIST assessed by investigate.
Objective Response Rate (ORR) ,Based on mRECIST | From the first dose of study drug to the first date of documentation of disease progression or death whichever occurred first (up to approximately 2 years )
  ORR was defined as the percentage of participants who had best overall response (BOR) of complete response (CR) or partial response (PR) based on mRECIST) assessed by investigator analysis.
Safety as measured by number and grade of adverse events | From first dose until 30 days after the last dose (up to approximately 2 years )
  Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: xuehao wang, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No